CLINICAL TRIAL: NCT03616912
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Study of Baricitinib in Patients With Systemic Lupus Erythematosus
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Systemic Lupus Erythematosus
Acronym: SLE-BRAVE I
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to insufficient evidence to support a positive benefit: risk profile in systemic lupus erythematosus patients.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16676; I4V-MC-JAHZ (Other: Eli Lilly and Company); 2017-005026-37 (EudraCT Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Participants received two placebo tablets: one matching baricitinib 4 milligram (mg) and one matching baricitinib 2 mg administered orally every day (QD) for 52 weeks.
  Interventions: Drug: Placebo
- 2 mg Baricitinib (Experimental): Participants received one Baricitinib 2 mg tablet and one placebo tablet matching Baricitinib 4 mg administered QD for 52 weeks.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 4 mg Baricitinib (Experimental): Participants received one Baricitinib 4 mg tablet and one placebo tablet matching baricitinib 2 mg administered orally every day (QD) for 52 weeks.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo Maximum Extended Enrollment (MEE) (Placebo Comparator): Participants received two placebo tablets: one matching baricitinib 4 mg and one matching baricitinib 2 mg administered orally QD for 52 weeks.
  Interventions: Drug: Placebo
- 2 mg Baricitinib (MEE) (Experimental): Participants received one Baricitinib 2 mg tablet and 1 placebo tablet matching Baricitinib 4 mg administered QD for 52 weeks.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 4 mg Baricitinib (MEE) (Experimental): Participants received one Baricitinib 4 mg tablet and one placebo tablet matching baricitinib 2 mg administered orally every day (QD) for 52 weeks.
  Interventions: Drug: Baricitinib; Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: 2 mg Baricitinib; 2 mg Baricitinib (MEE); 4 mg Baricitinib; 4 mg Baricitinib (MEE)
Drug: Placebo — Administered orally.

SUMMARY:
The reason for this study is to see how effective and safe the study drug known as baricitinib is in participants with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of SLE at least 24 weeks prior to screening.
* Have documentation of having met at least 4 of 11 Revised Criteria for Classification of Systemic Lupus Erythematosus according to the 1997 Update of the 1982 American College of Rheumatology (ACR) criteria for classification of SLE prior to randomization.
* Have a positive antinuclear antibody (ANA) (titer ≥1:80) and/or a positive anti-double-stranded deoxyribonucleic acid (dsDNA), and/or a positive anti-Smith (anti-Sm) as assessed by a central laboratory during screening.
* Have a total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥6 during screening.
* Have a clinical SLEDAI-2K score ≥4 at randomization.
* Have at least 1 British Isles Lupus Assessment Group (BILAG) A score or 2 BILAG B scores during screening.
* Are receiving at least one of the following standard of care medications for SLE:

  * A single antimalarial at a stable dose for at least 8 weeks prior to screening
  * A single immunosuppressant at a stable dose for at least 8 weeks prior to screening
  * An oral corticosteroid, initiated at least 4 weeks prior to screening, at a stable dose ≤40 milligrams/day prednisone (or equivalent) for at least 2 weeks prior to screening. If the participant is not receiving an antimalarial or immunosuppressant, the dose of corticosteroid must be ≥7.5 milligrams/day prednisone (or equivalent)

Exclusion Criteria:

* Have severe active lupus nephritis.
* Have active central nervous system (CNS) lupus.
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection.
* Have received cyclophosphamide (or any other cytotoxic agent) within 12 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (184):
- United States (60):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - University of Arizona, Tucson, Arizona
  - St. Joseph Heritage Medical Group, Fullerton, California
  - MD Medical Corporation, Hemet, California
  - ACRC Studies, Poway, California
  - Office: Hans R Barthel M.D., Santa Barbara, California
  - Medvin Clinical Research - Weidmann, Whittier, California
  - Denver Arthritis Clinic - Lowry, Denver, Colorado
  - New England Research Associates, Bridgeport, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Arthritis and Rheumatic Disease, Aventura, Florida
  - Rheumatology Associates of South Florida, Boca Raton, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Arthritis and Rheumatology Center of South Florida, Margate, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Millennium Research, Ormond Beach, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Atlanta Center for Clinical Research, Atlanta, Georgia
  - St Luke's Clinic - Intermountain Orthopaedics, Boise, Idaho
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - St. Louis Rheumatology, St Louis, Missouri
  - Glacier View Research Institute - Endocrinology, Kalispell, Montana
  - Allied Clinical Research, Reno, Nevada
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - SUNY Health Science Center, Brooklyn, New York
  - St. Lawrence Health System, Canton, New York
  - Northwell Health, Great Neck, New York
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Buffalo Rheumatology, Orchard Park, New York
  - Joint and Muscle Medical Care, Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Cincinnati Arthritis Associates, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Arthritis & Rheumatology Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - UPMC Lupus Center of Excellence, Pittsburgh, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Accurate Clinical Management, Baytown, Texas
  - Dr. Dhiman Basu Private Practice, Colleyville, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Precision Comprehensive Clinical Research Solutions, Fort Worth, Texas
  - Rheumatology Center of Houston, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Southwest Rheumatology, P.A., Mesquite, Texas
  - Accurate Clinical Research, Inc., San Antonio, Texas
  - Univ of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Arthritis Clinic Of Central Texas, San Marcos, Texas
  - Spectrum Medical Inc., Danville, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
- Australia (6):
  - Emeritus Research, Botany, New South Wales
  - The Rheumatology Research Unit Sunshine Coast, Maroochydore, Queensland
  - Emeritus Research, Camberwell, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Griffith University, Southport
- Austria (3):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Medizinische Universität Graz, Graz
  - Klinik Hietzing, Vienna
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - UZ Leuven, Leuven, Vlaams Brabant
  - CHU de Liège, Liège
- Brazil (10):
  - SER - Serviços Especializados em Reumatologia da Bahia S/S - ME, Salvador, Estado de Bahia
  - CIP-Centro Internacional de Pesquisa, Goiânia, Goiás
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras-CETI, Curitiba, Paraná
  - EDUMED - Educação em Saúde Ltda., Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - LMK Serviços Médicos S/S, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas UNICAMP, Campinas, São Paulo
  - Oncovida- Centro de Onco-Hematologia de Mato Grosso, Cuiabá
  - Hospital Alemao Oswaldo Cruz, São Paulo
- China (17):
  - The First Affliated Hospital of Soochow University, Suzhou, China
  - First affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of the Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou Universtiy, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Peking University First Hospital, Beijing
  - Beijing Peking Union Medical College Hospital, Beijing
  - Shanghai Huashan Hospital Affil to Fu Dan University, Shanghai
  - China Medical University (CMU) - First Affiliated Hospital, Shenyang
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi
- Croatia (3):
  - Klinicki Bolnicki Centar Rijeka, Rijeka
  - University Hospital Split, Split
  - Clinical Hospital Dubrava, Zagreb
- Czechia (5):
  - Revmatologicky ustav, Prague, Praha, Hlavní Mešto
  - Revmatologie.s.r.o., Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - ARTHROHELP s.r.o., Pardubice
  - Vseobecna fakultni nemocnice, Prague
- Germany (11):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Universitätsklinikum Würzburg A. ö. R., Würzburg, Bavaria
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universität Leipzig - Universitätsklinikum, Leipzig, Saxony
  - Charité Universitätsmedizin Berlin Campus Buch, Berlin
  - Immanuel Krankenhaus Rheuma Klinik Berlin Buch, Berlin
  - Schlosspark Klinik, Berlin
- Greece (5):
  - Gen Hospital of Athens G Gennimatas, Athens, Attica
  - University General Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Larissa, Larissa
  - Euromedica Kyanous Stavros General Hospital, Thessaloniki
  - Hippokration University Hopsital, Thessaloniki
- Hungary (10):
  - Bekes Megyei Pandy Kalman Korhaz, Gyula, Bekes County
  - Vital Medical Center, Veszprém, Veszprém City
  - Budai Irgalmasrendi Korhaz, Budapest
  - Qualiclinic Kft, Budapest
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointeze, Budapest
  - Debreceni Egyetem Klinikai Kozpont Reumatologiai Tanszek, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont I. Belgyogyaszati Klinika, Szeged
  - Vita Verum Egeszsegugyi Szolgaltato Bt, Székesfehérvár
- Israel (3):
  - Meir Medical Center, Kfar Saba
  - Chaim Sheba Medical Center, Ramat Gan
  - Carmel Hospital, Haifa, Ḥeifā
- Mexico (14):
  - CIMAB SA de CV, Torreón, Coahuila
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Guadalajara, Jalisco
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V., Zapopan, Jalisco
  - Cliditer Sa de CV, Mexico City, Mexico City
  - Hospital Angeles Lindavista, Mexico City, Mexico City
  - Centro Peninsular de Investigacion S.C.P, Mérida, Yucatán
  - Köhler & Milstein Research, Mérida, Yucatán
  - Cemdeicy S.C.P., Mérida, Yucatán
  - Clinosar Mexico S.A. de C.V, Mexico City
  - Centro de Investigación y Tratamiento Reumatológico S.C, Mexico City
  - Centro de Alta Especialidad Reumatologia e Inv Potosi, S.C., San Luis Potosí City
- Netherlands (2):
  - Medische Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Vrije Universiteit Medisch Centrum Amsterdam, Amsterdam
- Russia (16):
  - LLC MK Med, Saint Petersburg, Sankt-Peterburg
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - City Hospital # 7, Kazan'
  - Regional Clinical Hospital, Kursk
  - Russian State Medical University, Moscow
  - City Clinical Hospital 1 named after N.I. Pirogov, Moscow
  - Rheumatology Institute RAMS, Moscow
  - Healthy Family, Novosibirsk
  - Reafan, Novosibirsk
  - Institute of Cytology and Genetics of Siberian Branch of Russian Academy of Medical Sciences, Novosibirsk
  - Regional Hospital - Omsk, Omsk
  - Orenburg State Medical Academy of Roszdrav, Orenburg
  - Ryazan State Medical University, Ryazan
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Departmental Hospital at Smolensk Station "rzhd" JSC, Smolensk
  - Kuvatov Republican Clinical Hospital, Ufa
- Switzerland (2):
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
- Taiwan (9):
  - Chang Gung Memorial Hospital - Linkou, Kuei Shan Hsiang, Taoyuan Hsien
  - Hualien Tzu-Chi Hospital, Dalin Township
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
- United Kingdom (5):
  - Maidstone Hospital, Maidstone, Kent
  - Whipps Cross University Hospital, London, Surrey
  - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - Guy's Hospital, London
  - St. George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://trials.lillytrialguide.com/en-US/trial/64a5deI4M0sSScwYIMISsIDescriptionAStudyofBaricitinib(LY3009104)inParticipantsWithSystemicLupusErythematosus

REFERENCES:
- [Derived] Yin J, Hou Y, Wang C, Qin C. Clinical outcomes of baricitinib in patients with systemic lupus erythematosus: Pooled analysis of SLE-BRAVE-I and SLE-BRAVE-II trials. PLoS One. 2025 Apr 30;20(4):e0320179. doi: 10.1371/journal.pone.0320179. eCollection 2025. PMID 40305472
- [Derived] Morand EF, Vital EM, Petri M, van Vollenhoven R, Wallace DJ, Mosca M, Furie RA, Silk ME, Dickson CL, Meszaros G, Jia B, Crowe B, de la Torre I, Dorner T. Baricitinib for systemic lupus erythematosus: a double-blind, randomised, placebo-controlled, phase 3 trial (SLE-BRAVE-I). Lancet. 2023 Mar 25;401(10381):1001-1010. doi: 10.1016/S0140-6736(22)02607-1. Epub 2023 Feb 24. PMID 36848918
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: A Study of Baricitinib (LY3009104) in Participants With Systemic Lupus Erythematosus — https://trials.lillytrialguide.com/en-US/trial/64a5deI4M0sSScwYIMISsI

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One investigational site with seven participants was excluded from analysis due to confirmed misconduct.
Groups:
- 2 mg Baricitinib: Participants received one Baricitinib 2 mg tablet and one placebo tablet matching Baricitinib 4 mg administered orally QD for 52 weeks.
- 4 mg Baricitinib; 4 mg Baricitinib (MEE): Participants received one Baricitinib 4 mg tablet and one placebo tablet matching baricitinib 2 mg administered orally QD for 52 weeks.
- Placebo (MEE): Participants received two placebo tablets: one matching baricitinib 4 mg and one matching baricitinib 2 mg administered orally QD for 52 weeks.
- 2 mg Baricitinib (MEE): Participants received one Baricitinib 2 mg tablet and one placebo tablet matching Baricitinib 4 mg administered QD for 52 weeks.
Period: Overall Study
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib | Placebo (MEE) | 2 mg Baricitinib (MEE) | 4 mg Baricitinib (MEE)
Started | 257 | 258 | 254 | 21 | 20 | 20
Received at Least One Dose of Study Drug | 257 | 256 | 254 | 21 | 20 | 20
Excluded Due to Site Misconduct | 4 | 1 | 2 | 0 | 0 | 0
Completed | 204 | 211 | 208 | 5 | 5 | 6
Not Completed | 53 | 47 | 46 | 16 | 15 | 14
Not completed — Adverse Event | 17 | 21 | 9 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 13 | 6 | 8 | 4 | 5 | 1
Not completed — Lost to Follow-up | 1 | 2 | 3 | 0 | 0 | 0
Not completed — Due to Epidemic/Pandemic | 4 | 2 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 12 | 15 | 2 | 0 | 2
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 10 | 9 | 11
Not completed — Protocol Deviation | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Randomized But Never Treated | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who receive at least one dose of study drug. One investigational site with seven participants was excluded from analysis due to confirmed misconduct.
Groups:
- Placebo; Placebo Maximum Extended Enrollment (MEE): Participants received two placebo tablets: one matching baricitinib 4 mg and one matching baricitinib 2 mg administered orally QD for 52 weeks.
- 2 mg Baricitinib MEE: Participants received one Baricitinib 2 mg tablet and one placebo tablet matching Baricitinib 4 mg administered QD for 52 weeks.
- 4 mg Baricitinib MEE: Participants received one Baricitinib 4 mg tablet and one placebo tablet matching baricitinib 2 mg administered orally QD for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib | Placebo Maximum Extended Enrollment (MEE) | 2 mg Baricitinib MEE | 4 mg Baricitinib MEE | Total
Number analyzed (Participants) | 253 | 255 | 252 | 21 | 20 | 20 | 821
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.00 (11.98) | 42.90 (12.44) | 41.50 (12.88) | 32.90 (10.83) | 37.70 (11.38) | 34.60 (8.31) | 41.60 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 238 | 237 | 20 | 19 | 20 | 771
  Male | 16 | 17 | 15 | 1 | 1 | 0 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 13 | 11 | 0 | 0 | 0 | 28
  Not Hispanic or Latino | 42 | 35 | 38 | 0 | 0 | 0 | 115
  Unknown or Not Reported | 207 | 207 | 203 | 21 | 20 | 20 | 678
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 15 | 7 | 0 | 0 | 0 | 34
  Asian | 33 | 39 | 34 | 21 | 20 | 20 | 167
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 36 | 23 | 30 | 0 | 0 | 0 | 89
  White | 168 | 172 | 177 | 0 | 0 | 0 | 517
  More than one race | 1 | 2 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 3 | 4 | 4 | 0 | 0 | 0 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 10 | 9 | 12 | 0 | 0 | 0 | 31
  Austria | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Belgium | 2 | 1 | 1 | 0 | 0 | 0 | 4
  Brazil | 38 | 22 | 23 | 0 | 0 | 0 | 83
  China | 16 | 21 | 18 | 21 | 20 | 20 | 116
  Croatia | 5 | 3 | 2 | 0 | 0 | 0 | 10
  Czechia | 18 | 11 | 9 | 0 | 0 | 0 | 38
  Germany | 14 | 14 | 17 | 0 | 0 | 0 | 45
  Greece | 4 | 9 | 5 | 0 | 0 | 0 | 18
  Hungary | 13 | 18 | 19 | 0 | 0 | 0 | 50
  Israel | 1 | 3 | 4 | 0 | 0 | 0 | 8
  Mexico | 36 | 51 | 49 | 0 | 0 | 0 | 136
  Netherlands | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Russia | 26 | 25 | 20 | 0 | 0 | 0 | 71
  Switzerland | 3 | 2 | 3 | 0 | 0 | 0 | 8
  Taiwan | 15 | 11 | 13 | 0 | 0 | 0 | 39
  United Kingdom | 5 | 4 | 4 | 0 | 0 | 0 | 13
  United States | 47 | 49 | 50 | 0 | 0 | 0 | 146

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Systemic Lupus Erythematosus Responder Index 4 (SRI-4) Response (4 mg Baricitinib)
Description: SRI-4 response defined as 1)greater than or equal to (>=) 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score 2)no new British Isles Lupus Assessment Group (BILAG) A and no more than 1 new BILAG B domain score and 3)no worsening in Physician Global Assessment (PGA) of Disease Activity (worsening defined as an increase of >=0.3 from baseline on a 0-3 visual analogue scale).
  SLEDAI-2K assessment consists of 24 items with total score of 0(no symptoms) to 105 (presence of all defined symptoms) with higher scores representing increased disease activity. BILAG Index: assessing clinical signs, symptoms,or laboratory parameters related to Systemic Lupus Erythematosus (SLE),divided into 9 organ systems. For each organ system A=severe disease,B=moderate disease,C=mild stable disease,D=inactive,but previously active,E=inactive and never affected. PGA assess disease activity on a visual analogue scale from 0 to 3 (1=mild, 2=moderate, 3=severe).
Time Frame: Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (Modified intent to treat (mITT population). Missing data was imputed using the hybrid imputation method [nonresponder imputation (NRI) + multiple imputation (MI)]. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 4 mg Baricitinib
Number analyzed (Participants) | 253 | 252
percentage of participants | 45.9 | 56.7
Statistical Analysis 1: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.016, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [1.09 to 2.27]

2. Secondary Outcome: Percentage of Participants Achieving SRI-4 Response - 2 mg Baricitinib
Description: as for outcome 1
Time Frame: Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population). Missing data was imputed using the hybrid imputation method [nonresponder imputation (NRI) + multiple imputation (MI)]. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib
Number analyzed (Participants) | 253 | 255
percentage of participants | 45.9 | 49.8
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.470, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.79 to 1.65]

3. Secondary Outcome: Percentage of Participants Achieving a Lupus Low Disease Activity State (LLDAS)
Description: The LLDAS is a composite measure designed to identify patients achieving a state of low disease activity. The LLDAS response criteria were: (1) SLEDAI-2K <=4, with no activity in major organ systems (CNS, vascular, renal, cardiorespiratory and constitutional); where "no activity" is defined as all items of SLEDAI-2K within these major organ systems equal to 0. (2) no new features of lupus disease activity compared to previous occurred visit, where the "new feature" is defined as any of the SLEDAI-2K 24 items changed from 0 to greater than 0; (3) PGA (scale 0-3), <=1; (4) current prednisolone (or equivalent) dose <=7.5 mg daily.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 253 | 255 | 252
percentage of participants | 26.2 | 25.7 | 29.7
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.839, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.63 to 1.45]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.391, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.80 to 1.79]

4. Secondary Outcome: Time to First Severe Flare
Description: Time to first severe flare was analyzed using a Cox proportional hazards model with treatment group, baseline disease activity (Systemic Lupus Erythematosus Disease Activity Index 2000 [SLEDAI-2K ] <10; SLEDAI-2K ≥10), baseline corticosteroid dose (<10 mg/day; ≥10 mg/day prednisone or equivalent), and region fitted as explanatory variables. Participants who did not have severe flare during the flare exposure time period were censored at the end of the flare exposure time.
Time Frame: Baseline to Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population). As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 253 | 255 | 252
weeks | NA [NA to NA] — Data not available (NA) as < 50% of participants experienced first flare, median was not reached and 95% confidence interval could not be calculated. | NA [NA to NA] — Data not available (NA) as < 50% of participants experienced first flare, median was not reached and 95% confidence interval could not be calculated. | NA [NA to NA] — Data not available (NA) as < 50% of participants experienced first flare, median was not reached and 95% confidence interval could not be calculated.

5. Secondary Outcome: Percentage of Participants Whose Average Prednisone Dose Had Been Reduced by >=25% From Baseline to <=7.5 mg/Day During Weeks 40 Through 52 in Participants Receiving Greater Than 7.5 mg/Day at Baseline
Description: For the analysis of steroid use, steroid dosages were converted to a prednisone equivalent in mg. A responder was defined as having a prednisone reduction by >=25% from Baseline to <=7.5 mg/day during Weeks 40 through 52.
Time Frame: Baseline, Week 40 through Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population) and received >7.5 mg prednisone at baseline. Missing data was imputed using the hybrid imputation method [NRI + modified last observation carried forward]. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 117 | 106 | 106
percentage of participants | 30.8 | 29.2 | 34.0
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.820, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.53 to 1.66]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.565, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.67 to 2.08]

6. Secondary Outcome: Change From Baseline in Worst Pain Numeric Rating Scale (NRS)
Description: Participants assessed their worst pain in the last 24 hours on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The average worst daily pain score was calculated as the mean of the scores over the last 7 days prior to each assessment time point. Higher score indicated severe pain. Least Squares (LS) mean was calculated using Mixed Model Repeated Measures (MMRM) analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >= 10 mg/day prednisone or equivalent), region (North America, Central/South, America/Mexico, Europe, Asia Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population) and had baseline and post-baseline values at the specified time point. Missing data was imputed using the hybrid imputation method (NRI + MMRM). As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 173 | 173 | 182
score on a scale | -1.62 (0.15) | -1.73 (0.15) | -1.71 (0.15)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.598, Mixed Models Analysis; LS Mean Difference Final Values = -0.11, 95% CI 2-sided [-0.52 to 0.30], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.674, Mixed Models Analysis; LS Mean Difference Final Values = -0.09, 95% CI 2-sided [-0.50 to 0.32], Standard Error of Mean 0.21

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Total Score
Description: FACIT-Fatigue score calculated according to a 13-item questionnaire that assess self reported fatigue and its impact upon daily activities and function. It uses a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse possible score) to 52 (best score). A higher score reflected an improvement in the participant's health status. Least Squares (LS) mean was calculated using Mixed Model Repeated Measures (MMRM) analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >= 10 mg/day prednisone or equivalent), region (North America, Central/South, America/Mexico, Europe, Asia Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population) and had baseline and post-baseline values at the specified time-point. Missing data was imputed using the hybrid imputation method (NRI + MMRM). As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Participants received two placebo tablets: one matching baricitinib 4 mg and one matching baricitinib 2 mg administered orally every day QD for 52 weeks.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 188 | 201 | 204
score on a scale | 7.44 (0.62) | 7.46 (0.60) | 7.08 (0.61)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.979, Mixed Models Analysis; LS Mean Difference Final Values = 0.02, 95% CI 2-sided [-1.65 to 1.70], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.678, Mixed Models Analysis; LS Mean Difference Final Values = -0.36, 95% CI 2-sided [-2.03 to 1.32], Standard Error of Mean 0.86

8. Secondary Outcome: Percentage of Participants With Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Total Activity Score ≥10 at Baseline With ≥50% Reduction in CLASI Total Activity Score
Description: The CLASI is a single-page tool that separately quantifies disease activity and damage. For the activity score, points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. The total score represents the sum of the individual scores and ranges from 0 to 70. Higher scores are awarded for more severe manifestations.
Time Frame: Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population) and had baseline CLASI score of >= 10. Missing data was imputed using NRI method. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 49 | 46 | 43
percentage of participants | 49.0 | 54.3 | 55.8
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.965, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.43 to 2.42]
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.661, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.51 to 2.92]

9. Secondary Outcome: Change From Baseline in Tender Joints Count
Description: The number of tender and painful joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as tender or not tender. LS mean was calculated using Mixed Model Repeated Measures (MMRM) analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >=10 mg/day prednisone or equivalent), region (North America, Central/South America/Mexico, Europe, Asia and Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population) and had baseline and post-baseline values at specified time point. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: tender joint count
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 183 | 198 | 195
tender joint count | -7.50 (0.312) | -7.26 (0.305) | -7.94 (0.307)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.578, Mixed Models Analysis; LS Mean Difference Final Values = 0.24, 95% CI 2-sided [-0.61 to 1.08], Standard Error of Mean 0.430
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.309, Mixed Models Analysis; LS Mean Difference Final Values = -0.44, 95% CI 2-sided [-1.29 to 0.41], Standard Error of Mean 0.433

10. Secondary Outcome: Change From Baseline in Swollen Joint Count
Description: The number of swollen joints is determined by examination of 28 joints (14 on each side) which include: the 2 shoulders, the 2 elbows, the 2 wrists, the 10 metacarpophalangeal joints, the 2 interphalangeal joints of the thumb, the 8 proximal interphalangeal joints, and the 2 knees. The joints are assessed and classified as swollen or not swollen. LS mean was calculated using MMRM analysis with treatment, baseline disease activity (total SLEDAI-2K <10; >=10), baseline corticosteroid dose (<10 mg/day; >=10 mg/day prednisone or equivalent), region (North America, Central/South America/Mexico, Europe, Asia and Rest of World), visit (as categorical variable), baseline value, treatment-by-visit interaction, and baseline value-by-visit interaction.
Time Frame: Baseline, Week 52
Population: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug (mITT population) and had baseline and post-baseline values at the specified time point. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: swollen joint count
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 183 | 198 | 195
swollen joint count | -5.37 (0.201) | -5.67 (0.196) | -5.81 (0.198)
Statistical Analysis 1: Comparison: Placebo vs 2 mg Baricitinib; Test type: Superiority; p = 0.287, Mixed Models Analysis; LS Mean Difference Final Values = -0.29, 95% CI 2-sided [-0.84 to 0.25], Standard Error of Mean 0.277
Statistical Analysis 2: Comparison: Placebo vs 4 mg Baricitinib; Test type: Superiority; p = 0.113, Mixed Models Analysis; LS Mean Difference Final Values = -0.44, 95% CI 2-sided [-0.99 to 0.11], Standard Error of Mean 0.278

11. Secondary Outcome: Population Pharmacokinetics (PK): Area Under the Concentration-Time Curve of Baricitinib at Steady State (AUCτ, ss)
Description: PK: Area Under the Concentration-Time Curve of Baricitinib at Steady State (AUCτ, ss) was evaluated using population PK approach.
Time Frame: Week 0 (Baseline): 15 minutes (min) and 60 min postdose; Week 4: 2 to 4 hours (hr) postdose; Week 8: 4 to 6 hr postdose; Week 12 and Week 16 predose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data. As pre-specified in the analysis plan, outcome measures will not be reported for the MEE arms/groups but only for the main global study arms/groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter (h*ng/mL)
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 248 | 220
hour*nanograms per milliliter (h*ng/mL) | 256 (52) | 502 (52)

12. Secondary Outcome: Population PK: Maximum Observed Drug Concentration at Steady State (Cmax,ss)
Description: Population PK: Maximum Observed Drug Concentration at Steady State (Cmax,ss) was evaluated using population PK approach.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 2 mg Baricitinib | 4 mg Baricitinib
Number analyzed (Participants) | 248 | 220
nanograms per milliliter (ng/mL) | 26.7 (24) | 53.0 (23)

ADVERSE EVENTS:
Time Frame: Baseline through Follow-up (Up to 56 Weeks)
Description: All randomized participants, excluding participants from site with confirmed misconduct, who received at least one dose of study drug and who did not discontinue from the study for the reason "Lost to Follow-up" at the first postbaseline visit. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | 2 mg Baricitinib | 4 mg Baricitinib | Placebo Maximum Extended Enrollment (MEE) | 2 mg Baricitinib (MEE) | 4 mg Baricitinib (MEE)
All-Cause Mortality (participants affected / at risk) | 1/253 | 1/255 | 0/252 | 0/21 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 19/253 | 27/255 | 31/252 | 1/21 | 4/20 | 3/20
Other Adverse Events (participants affected / at risk) | 129/253 | 144/255 | 144/252 | 17/21 | 14/20 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=253) | 2 mg Baricitinib (N=255) | 4 mg Baricitinib (N=252) | Placebo Maximum Extended Enrollment (MEE) (N=21) | 2 mg Baricitinib (MEE) (N=20) | 4 mg Baricitinib (MEE) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0/237 (0) | 1/238 (1) | 0/237 (0) | 0/20 (0) | 0/19 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Device use issue (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/237 (1) | 0/238 (0) | 0/237 (0) | 0/20 (0) | 0/19 (0) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/237 (1) | 0/238 (0) | 1/237 (1) | 0/20 (0) | 0/19 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/237 (0) | 0/238 (0) | 1/237 (1) | 0/20 (0) | 0/19 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0/237 (0) | 0/238 (0) | 1/237 (1) | 0/20 (0) | 0/19 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/237 (0) | 0/238 (0) | 1/237 (1) | 0/20 (0) | 0/19 (0) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 0/237 (0) | 1/238 (1) | 0/237 (0) | 0/20 (0) | 0/19 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1/237 (1) | 0/238 (0) | 0/237 (0) | 0/20 (0) | 0/19 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=253) | 2 mg Baricitinib (N=255) | 4 mg Baricitinib (N=252) | Placebo Maximum Extended Enrollment (MEE) (N=21) | 2 mg Baricitinib (MEE) (N=20) | 4 mg Baricitinib (MEE) (N=20)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 4 (6) | 13 (16) | 3 (4) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 10 (13) | 11 (14) | 9 (10) | 3 (3) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 2 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 10 (12) | 10 (12) | 1 (1) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 11 (13) | 12 (14) | 0 (0) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 1 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (4) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Covid-19 (Infections and infestations) | 9 (9) | 16 (16) | 13 (13) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Herpes zoster (Infections and infestations) | 8 (8) | 9 (9) | 16 (18) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 17 (24) | 19 (21) | 18 (24) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 17 (19) | 21 (30) | 19 (27) | 5 (11) | 9 (17) | 7 (8)
Urinary tract infection (Infections and infestations) | 25 (38) | 32 (41) | 37 (47) | 2 (2) | 3 (3) | 1 (1)
Vulvitis (Infections and infestations) | 0/237 (0) | 0/238 (0) | 0/237 (0) | 0/20 (0) | 1/19 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 6 (8) | 2 (5) | 1 (1) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 3 (4) | 8 (9) | 14 (20) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Weight increased (Investigations) | 7 (9) | 5 (5) | 3 (3) | 2 (4) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 6 (6) | 3 (4) | 4 (4) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 (5) | 9 (9) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 2 (2) | 2 (3) | 3 (3) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 25 (26) | 16 (19) | 20 (23) | 1 (3) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (8) | 4 (4) | 5 (6) | 1 (1) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0/16 (0) | 1/17 (1) | 0/15 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 7 (7) | 2 (2) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 4 (4) | 2 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 10 (10) | 17 (18) | 17 (18) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
One investigational site with seven participants was excluded from analysis due to confirmed misconduct.

Study terminated due to insufficient evidence to support a positive benefit: risk profile in systemic lupus erythematosus patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03616912/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03616912/SAP_001.pdf